CLINICAL TRIAL: NCT03397316
Title: Evaluation of Marginal Bone Loss After Immediate Implant Placement in Maxillary Esthetic Zone With and Without Xenograft.
Brief Title: Evaluation of Marginal Bone Loss After Immediate Implant Placement in Esthetic Zone Without Xenograft.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Alaa Eldin Mohamed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AlaaCUImplant
Record Dates: First submitted 2018-01-01; First posted 2018-01-12 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Bone Loss
Keywords: immediate implant; upper esthetic zone; marginal bone loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each patient will be given a code by researcher (A.A) and the observers will be blind to which group this case belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Marginal bone loss without grafting. (No Intervention): immediate implant placement in upper esthetic zone.
- marginal bone loss with xenograft. (Active Comparator): xenograft placement (Geistlich Bio-Oss) in immediate implant placement in upper esthetic zone between the residual labial bone and implant surface.
  Interventions: Procedure: xenograft placement .

INTERVENTIONS:
Procedure: xenograft placement . — immediate implant placement in upper esthetic zone with xenograft placement between residual labial bone and implant surface.
  Arms: marginal bone loss with xenograft.

SUMMARY:
Marginal bone loss in immediate implant placement in upper esthetic zone by comparing between non grafting in immediate implant placement with xenograft placement in other side.

the study is to assess the marginal bone loss in the two techniques and compare results between them.

DETAILED DESCRIPTION:
Marginal bone loss in immediate implant placement in upper esthetic zone by comparing between non grafting in immediate implant placement with xenograft placement in other side.

the study is to assess the marginal bone loss in the two techniques and compare results between them after follow up period of 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with badly broken teeth in upper esthetic zone indicated for extraction presence of at least 4 mm of bone beyond root apex

Exclusion Criteria:

* presence of fenestrations or dehiscences of the residual bony walls after extraction heavy smokers more than 20 cigarettes per day. systemic diseases that may affect normal healing. psychiatric problems.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-15 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
marginal bone loss | 4 months
  Evaluation of marginal bone loss after Immediate implant placement in maxillary esthetic zone with and without xenograft

SECONDARY OUTCOMES:
patient satisfaction | 4 months
  measure patient satisfaction by patient satisfaction chart.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided